CLINICAL TRIAL: NCT06005597
Title: A Placebo-Controlled, Double-Blind, Randomized, Phase 3 Study to Evaluate the Effect of Obicetrapib 10 mg and Ezetimibe 10 mg Fixed Dose Combination Daily on Top of Maximally Tolerated Lipid-Modifying Therapy in Participants With Heterozygous Familial Hypercholesterolemia (HeFH) and/or Atherosclerotic Cardiovascular Disease (ASCVD) or Multiple ASCVD Risk Factors
Brief Title: Study of Obicetrapib & Ezetimibe Fixed Dose Combination on Top of Maximum Tolerated Lipid-Modifying Therapies
Acronym: TANDEM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NewAmsterdam Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OBEZ-301
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Results first posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Dyslipidemias; Hypercholesterolemia; Familial Hypercholesterolemia; ASCVD; High Cholesterol
Keywords: obicetrapib; statin; LDL-C; cholesterol; atherosclerosis
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia; Hyperlipoproteinemia Type II; Atherosclerosis | interventions — Combined Modality Therapy; Cholesterol Ester Transfer Proteins; Ezetimibe

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, double blind, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo tablets made to resemble active; placebo capsule made to resemble active
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Combination Therapy (Experimental): once-daily obicetrapib 10 mg and ezetimibe 10 mg fixed dose combination tablet, placebo tablet, placebo capsule
  Interventions: Combination Product: Combination Therapy; Other: Obicetrapib Placebo; Other: Ezetimibe Placebo
- Monotherapy obicetrapib (Experimental): once-daily obicetrapib 10 mg, placebo tablet, placebo capsule
  Interventions: Drug: Monotherapy obicetrapib; Other: Combination Therapy placebo; Other: Ezetimibe Placebo
- Monotherapy ezetimibe (Active Comparator): once-daily ezetimibe 10 mg capsule, 2 placebo tablets
  Interventions: Drug: Monotherapy ezetimibe; Other: Combination Therapy placebo; Other: Obicetrapib Placebo
- Placebo (Placebo Comparator): once-daily placebo tablets (2), placebo capsule
  Interventions: Other: Combination Therapy placebo; Other: Obicetrapib Placebo; Other: Ezetimibe Placebo

INTERVENTIONS:
Combination Product: Combination Therapy — tablet; 10mg obicetrapib and 10mg ezetimibe fixed does combination
  Other Names: Cholesteryl ester transfer protein (CETP) inhibitor; obicetrapib; ezetimibe
  Arms: Combination Therapy
Drug: Monotherapy obicetrapib — tablet; 10mg obicetrapib
  Other Names: CETP inhibitor
  Arms: Monotherapy obicetrapib
Drug: Monotherapy ezetimibe — capsule; 10mg ezetimibe
  Arms: Monotherapy ezetimibe
Other: Combination Therapy placebo — tablet; no active ingredient
  Arms: Monotherapy ezetimibe; Monotherapy obicetrapib; Placebo
Other: Obicetrapib Placebo — tablet; no active ingredient
  Arms: Combination Therapy; Monotherapy ezetimibe; Placebo
Other: Ezetimibe Placebo — capsule; no active ingredient
  Arms: Combination Therapy; Monotherapy obicetrapib; Placebo

SUMMARY:
The study is a placebo-controlled, double-blind, randomized, phase 3 study in participants with heterozygous familial hypercholesterolemia (HeFH) and/or atherosclerotic cardiovascular disease (ASCVD) or multiple ASCVD risk factors to evaluate the efficacy, safety and tolerability of obicetrapib 10mg and ezetimibe 10mg fixed dose combination as an adjunct to diet and maximally tolerated lipid-lowering therapy.

DETAILED DESCRIPTION:
This study will be a placebo-controlled, double-blind, randomized, phase 3 study in participants with heterozygous familial hypercholesterolemia (HeFH) and/or atherosclerotic cardiovascular disease (ASCVD) or multiple ASCVD risk factors to evaluate the efficacy, safety, and tolerability of obicetrapib as an adjunct to diet and maximally tolerated lipid-lowering therapy. The screening period for this study will take up to 14 days. Afterwards patients will be randomized 1:1:1:1 to Obicetrapib 10 mg and ezetimibe 10 mg fixed dose combination, obicetrapib 10 mg, ezetimibe 10 mg or placebo for a 84 day treatment period. After the treatment period, patients will have an end of study follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Have underlying HeFH and/or a history of ASCVD or multiple ASCVD risk factors
* On maximally tolerated lipid-modifying therapy as an adjunct to a diet and lifestyle modifications
* LDL-C ≥ 70 mg/dL
* Triglycerides < 500
* Estimated glomerular filtration rate ≥ 15 mL/min/1.73 m2

Exclusion Criteria:

* History of New York Heart Association (NYHA) class III or IV heart failure of left ventricular ejection fraction <30%
* Hospitalized for heart failure within the last 5 years
* Myocardial infarction, stroke, non-elective coronary revascularization or hospitalization for unstable angina or chest pain in the last 3 months
* Uncontrolled severe hypertension
* Diagnosis of homozygous FH
* Liver disease
* HbA1c ≥ 10.0% or fasting glucose ≥ 270 mg/dL
* Thyroid-stimulating hormone >1.5 x upper limit of normal (ULN)
* History of malignancy
* Creatinine kinase (CK) >3 X ULN
* Alcohol abuse
* Treatment with investigational product
* Treatment with gemfibrozil or ezetimibe
* Previous participation in a trial evaluating obicetrapib
* Known allergy to study drugs, placebo or excipients in study drugs of placebo
* Other condition that would interfere with the conduct of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ditmarsch, MD, Study Director — NewAmsterdam Pharma
Locations (45):
- United States (45):
  - East Valley Diabetes & Endocrinology, Gilbert, Arizona
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Centricity Research - Columbus, Columbus, Georgia
  - Center for Advanced Research and Education, Gainesville, Georgia
  - NSC Research, Johns Creek, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Evanston Premier Healthcare Research LLC, Skokie, Illinois
  - Cardiovascular Research of Northwest Indiana, LLC, Munster, Indiana
  - Grace Research, LLC - Bossier City, LA, Bossier City, Louisiana
  - Horizon Research Group of Opelousas, Eunice, Louisiana
  - Maryland Cardiovascular Specialists, Baltimore, Maryland
  - TidalHealth Peninsula Regional, Inc., Salisbury, Maryland
  - McClaren Bay Heart and Vascular, Bay City, Michigan
  - Northern Pines Health Center, Buckley, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Oakland Medical Research Center, Troy, Michigan
  - CentraCare Heart & Vascular Center, Saint Cloud, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - St. Louis Heart and Vascular Cardiology, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Triad Internal Medicine, Asheboro, North Carolina
  - Cary Research Group, LLC, Cary, North Carolina
  - Novant Health Clinical Research, LLC, Charlotte, North Carolina
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - Lucas Research, Inc, Morehead City, North Carolina
  - Wilmington Health Associates, Wilmington, North Carolina
  - Metabolic and Atherosclerosis Research Center, Cincinnati, Ohio
  - Summit Research Group, LLC, Stow, Ohio
  - Capital Area Research, Camp Hill, Pennsylvania
  - Monument Health Clinical Research, a department of Monument Health Rapid City Hospital, Inc, Rapid City, South Dakota
  - Chattanooga Research & Medicine, PLLC, Chattanooga, Tennessee
  - Cardiovascular Research of Knoxville, Powell, Tennessee
  - PharmaTex Research, LLC, Amarillo, Texas
  - Amarillo Heart Clinical Research Institute, Inc, Amarillo, Texas
  - South Texas Clinical Research, Corpus Christi, Texas
  - Diabetes and Thyroid Center of Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Juno Research, LLC - Medical Center Office, Houston, Texas
  - DM Clinical Research, Houston, Texas
  - Wellness Clinical Research Associates, McKinney, Texas
  - Northwest Houston Heart Center, Tomball, Texas
  - Alpine Research Organization, Inc., Clinton, Utah
  - Spectrum Medical, Inc., Danville, Virginia
  - Hampton Roads Center for Clinical Research, Suffolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sarraju A, Brennan D, Hayden K, Stronczek A, Goldberg AC, Michos ED, McGuire DK, Mason D, Tercek G, Nicholls SJ, Kling D, Neild AL, Kastelein J, Davidson M, Ditmarsch M, Nissen SE. Fixed-dose combination of obicetrapib and ezetimibe for LDL cholesterol reduction (TANDEM): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet. 2025 May 17;405(10491):1757-1768. doi: 10.1016/S0140-6736(25)00721-4. Epub 2025 May 7. PMID 40347969
- See also: Study results paper — https://pubmed.ncbi.nlm.nih.gov/40347969/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 716 participants were screened: out of 716, 407 participants were randomized (1:1:1:1) (FDC therapy: Obicetrapib monotherapy: Ezetimibe monotherapy: placebo)
Groups:
- Fixed Dose Combination: once-daily obicetrapib 10 mg and ezetimibe 10 mg fixed dose combination tablet, placebo tablet, placebo capsule
  Fixed Dose Combination: tablet; 10mg obicetrapib and 10mg ezetimibe fixed does combination
  Obicetrapib Placebo: tablet; no active ingredient
  Ezetimibe Placebo: capsule; no active ingredient
Period: Overall Study
Arm/Group | Fixed Dose Combination | Monotherapy Obicetrapib | Monotherapy Ezetimibe | Placebo
Started | 102 | 102 | 101 | 102
Completed | 100 | 99 | 99 | 100
Not Completed | 2 | 3 | 2 | 2
Not completed — Lost to Follow-up | 1 | 2 | 1 | 2
Not completed — Death | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Population is defined as all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed Dose Combination | Monotherapy Obicetrapib | Monotherapy Ezetimibe | Placebo | Total
Number analyzed (Participants) | 102 | 102 | 101 | 102 | 407
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (9.43) | 66.7 (9.64) | 67.6 (8.71) | 66.1 (9.47) | 66.9 (9.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 33 | 45 | 51 | 177
  Male | 54 | 69 | 56 | 51 | 230
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 1 | 2 | 9
  Not Hispanic or Latino | 98 | 100 | 100 | 100 | 398
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 2
  Asian | 1 | 0 | 3 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 14 | 15 | 13 | 17 | 59
  White | 86 | 85 | 82 | 84 | 337
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 0 | 3
Baseline Low-Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] — Baseline LDL-C is defined as the last measurement prior to the first dose of study drug. LDL-C was measured by Preparative Ultracentrifugation (PUC).
  mg/dL | 96.5 (28.80) | 100.0 (35.34) | 98.2 (31.09) | 91.0 (25.81) | 96.4 (30.26)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Fixed-Dose Combination (FDC) Compared to Placebo on LDL-C
Description: LS mean percent change in low-density lipoprotein cholesterol (LDL-C) from baseline to Day 84 in the obicetrapib 10 mg/ezetimibe 10 mg fixed-dose combination (FDC) group compared to the placebo group. LDL-C level was measured by preparative ultracentrifugation (PUC).
Time Frame: 84 Days
Population: Baseline Population is defined as all participants who were randomized in the study. Baseline values were defined as last measurement prior to the first dose of study drug. Missing values were imputed using a multiple imputation model assuming the data were missing not at random. Missing measurements of non-retrieved dropouts were modeled by known measurements from retrieved dropouts in the same treatment group.
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Groups:
- Fixed Dose Combination: once-daily obicetrapib 10 mg and ezetimibe 10 mg fixed dose combination tablet, placebo tablet, placebo capsule
  Fixed Dose Combination: tablet; 10 mg obicetrapib and 10 mg ezetimibe fixed does combination
  Obicetrapib Placebo: tablet; no active ingredient
  Ezetimibe Placebo: capsule; no active ingredient
Arm/Group | Fixed Dose Combination | Placebo
Number analyzed (Participants) | 102 | 100
percent change from baseline | -45.58 (3.465) | 3.03 (3.564)
Statistical Analysis 1: Comparison: Fixed Dose Combination vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -48.61, 95% CI 2-sided [-58.33 to -38.89], Standard Error of Mean 4.959

2. Primary Outcome: Effect of Fixed Dose Combination (FDC) Compared to Ezetimibe Monotherapy on LDL-C
Description: LS mean percent change in low-density lipoprotein cholesterol (LDL-C) from baseline to Day 84 in the obicetrapib 10 mg/ezetimibe 10 mg fixed-dose combination (FDC) group compared to the ezetimibe monotherapy 10 mg group. LDL-C level was measured by preparative ultracentrifugation (PUC).
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Fixed Dose Combination | Monotherapy Ezetimibe
Number analyzed (Participants) | 102 | 101
percent change from baseline | -45.58 (3.465) | -17.63 (3.497)
Statistical Analysis 1: Comparison: Fixed Dose Combination vs Monotherapy Ezetimibe; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -27.94, 95% CI 2-sided [-37.53 to -18.35], Standard Error of Mean 4.893

3. Primary Outcome: Effect of Fixed Dose Combination (FDC) Compared to Obicetrapib Monotherapy on LDL-C
Description: LS mean percent change in low-density lipoprotein cholesterol (LDL-C) from baseline to Day 84 in the obicetrapib 10 mg/ezetimibe 10 mg fixed-dose combination (FDC) group compared to the obicetrapib monotherapy 10 mg group. LDL-C level was measured by preparative ultracentrifugation (PUC).
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Groups:
- Fixed Dose Combination: once-daily obicetrapib 10 mg and ezetimibe 10 mg fixed dose combination tablet, placebo tablet, placebo capsule
  Fixed Dose Combination: tablet; 10 mg obicetrapib and 10mg ezetimibe fixed does combination
  Obicetrapib Placebo: tablet; no active ingredient
  Ezetimibe Placebo: capsule; no active ingredient
- Monotherapy Obicetrapib: once-daily obicetrapib 10 mg, placebo tablet, placebo capsule
  Monotherapy obicetrapib: tablet; 10 mg obicetrapib
  Combination Therapy placebo: tablet; no active ingredient
  Ezetimibe Placebo: capsule; no active ingredient
Arm/Group | Fixed Dose Combination | Monotherapy Obicetrapib
Number analyzed (Participants) | 102 | 102
percent change from baseline | -45.58 (3.465) | -28.82 (3.484)
Statistical Analysis 1: Comparison: Fixed Dose Combination vs Monotherapy Obicetrapib; Test type: Superiority; p = 0.0007, ANCOVA; Least Squares (LS) Means = -16.76, 95% CI 2-sided [-26.40 to -7.12], Standard Error of Mean 4.918

4. Primary Outcome: Effect of Obicetrapib Monotherapy Compared to Placebo on LDL-C
Description: LS mean percent change in low-density lipoprotein cholesterol (LDL-C) from baseline to Day 84 in the obicetrapib 10 mg group compared to the placebo group. LDL-C level was measured by preparative ultracentrifugation (PUC).
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Monotherapy Obicetrapib | Placebo
Number analyzed (Participants) | 102 | 100
percent change from baseline | -28.82 (3.484) | 3.03 (3.564)
Statistical Analysis 1: Comparison: Monotherapy Obicetrapib vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -31.85, 95% CI 2-sided [-41.64 to -22.07], Standard Error of Mean 4.993

5. Secondary Outcome: Effect of Fixed Dose Combination (FDC) Compared to Placebo on Non-HDL-C
Description: LS mean percent change in non-high-density lipoprotein cholesterol (Non-HDL-C) from baseline to Day 84 in the obicetrapib 10 mg/ezetimibe 10 mg fixed-dose combination (FDC) group compared to the placebo group.
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Fixed Dose Combination | Placebo
Number analyzed (Participants) | 102 | 102
percent change from baseline | -42.42 (2.977) | 2.71 (3.017)
Statistical Analysis 1: Comparison: Fixed Dose Combination vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -45.13, 95% CI 2-sided [-53.43 to -36.84], Standard Error of Mean 4.233

6. Secondary Outcome: Effect of Fixed Dose Combination (FDC) Compared to Placebo on Apolipoprotein B (ApoB)
Description: LS mean percent change in apolipoprotein B (ApoB) from baseline to Day 84 in the obicetrapib 10 mg/ezetimibe 10 mg fixed-dose combination (FDC) group compared to the placebo group.
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Fixed Dose Combination | Placebo
Number analyzed (Participants) | 102 | 102
percent change from baseline | -26.91 (2.425) | 2.28 (2.466)
Statistical Analysis 1: Comparison: Fixed Dose Combination vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -29.19, 95% CI 2-sided [-35.99 to -22.40], Standard Error of Mean 3.467

7. Secondary Outcome: Effect of Obicetrapib Monotherapy Compared to Placebo on Non-HDL-C
Description: LS mean percent change in non-high-density lipoprotein cholesterol (Non-HDL-C) from baseline to Day 84 in the obicetrapib monotherapy 10 mg group compared to the placebo group.
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Monotherapy Obicetrapib | Placebo
Number analyzed (Participants) | 102 | 102
percent change from baseline | -27.19 (3.010) | 2.71 (3.017)
Statistical Analysis 1: Comparison: Monotherapy Obicetrapib vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -29.90, 95% CI 2-sided [-38.28 to -21.53], Standard Error of Mean 4.274

8. Secondary Outcome: Effect of Obicetrapib Monotherapy Compared to Placebo on Apolipoprotein B (ApoB)
Description: LS mean percent change in apolipoprotein B (ApoB) from baseline to Day 84 in the obicetrapib monotherapy 10 mg group compared to the placebo group.
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Monotherapy Obicetrapib | Placebo
Number analyzed (Participants) | 102 | 102
percent change from baseline | -17.50 (2.482) | 2.28 (2.466)
Statistical Analysis 1: Comparison: Monotherapy Obicetrapib vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -19.78, 95% CI 2-sided [-26.73 to -12.82], Standard Error of Mean 3.549

9. Secondary Outcome: Effect of Fixed-Dose Combination (FDC) Compared to Ezetimibe Monotherapy on Non-HDL-C
Description: LS mean percent change in non-high-density lipoprotein cholesterol (Non-HDL-C) from baseline to Day 84 in the obicetrapib 10 mg/ezetimibe 10 mg fixed-dose combination (FDC) group compared to the ezetimibe monotherapy 10 mg group.
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Groups:
- Monotherapy Ezetimibe: once-daily ezetimibe 10 mg capsule, 2 placebo tablets
  Monotherapy ezetimibe: capsule; 10 mg ezetimibe
  Combination Therapy placebo: tablet; no active ingredient
  Obicetrapib Placebo: tablet; no active ingredient
Arm/Group | Fixed Dose Combination | Monotherapy Ezetimibe
Number analyzed (Participants) | 102 | 101
percent change from baseline | -42.42 (2.977) | -16.98 (3.006)
Statistical Analysis 1: Comparison: Fixed Dose Combination vs Monotherapy Ezetimibe; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -25.44, 95% CI 2-sided [-33.67 to -17.22], Standard Error of Mean 4.198

10. Secondary Outcome: Effect of Fixed-Dose Combination (FDC) Compared to Ezetimibe Monotherapy on Apolipoprotein B (ApoB)
Description: LS mean percent change in apolipoprotein B (ApoB) from baseline to Day 84 in the obicetrapib 10 mg/ezetimibe 10 mg fixed-dose combination (FDC) group compared to the ezetimibe monotherapy 10 mg group.
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Fixed Dose Combination | Monotherapy Ezetimibe
Number analyzed (Participants) | 102 | 101
percent change from baseline | -26.91 (2.425) | -12.71 (2.495)
Statistical Analysis 1: Comparison: Fixed Dose Combination vs Monotherapy Ezetimibe; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -14.21, 95% CI 2-sided [-21.06 to -7.36], Standard Error of Mean 3.495

11. Secondary Outcome: Effect of Fixed-Dose Combination (FDC) Compared to Obicetrapib Monotherapy on Non-HDL-C
Description: LS mean percent change in non-high-density lipoprotein cholesterol (Non-HDL-C) from baseline to Day 84 in the obicetrapib 10 mg/ezetimibe 10 mg fixed-dose combination (FDC) group compared to the obicetrapib monotherapy 10mg group.
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Fixed Dose Combination | Monotherapy Obicetrapib
Number analyzed (Participants) | 102 | 102
percent change from baseline | -42.42 (2.977) | -27.19 (3.010)
Statistical Analysis 1: Comparison: Fixed Dose Combination vs Monotherapy Obicetrapib; Test type: Superiority; p = 0.0003, ANCOVA; Least Squares (LS) Means = -15.23, 95% CI 2-sided [-23.53 to -6.93], Standard Error of Mean 4.236

12. Secondary Outcome: Effect of Fixed-Dose Combination (FDC) Compared to Obicetrapib Monotherapy on Apolipoprotein B (ApoB)
Description: LS mean percent change in Apolipoprotein B (ApoB) from baseline to Day 84 in the obicetrapib 10 mg/ezetimibe 10 mg fixed-dose combination (FDC) group compared to the obicetrapib monotherapy 10 mg group.
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Fixed Dose Combination | Monotherapy Obicetrapib
Number analyzed (Participants) | 102 | 102
percent change from baseline | -26.91 (2.425) | -17.50 (2.482)
Statistical Analysis 1: Comparison: Fixed Dose Combination vs Monotherapy Obicetrapib; Test type: Superiority; p = 0.007, ANCOVA; Least Squares (LS) Means = -9.42, 95% CI 2-sided [-16.26 to -2.57], Standard Error of Mean 3.493

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 16
Description: Safety Population included all participants who received at least 1 dose of any study drug.
Arm/Group | Fixed Dose Combination | Monotherapy Obicetrapib | Monotherapy Ezetimibe | Placebo
All-Cause Mortality (participants affected / at risk) | 1/102 | 1/102 | 1/101 | 0/102
Serious Adverse Events (participants affected / at risk) | 3/102 | 6/102 | 7/101 | 4/102
Other Adverse Events (participants affected / at risk) | 30/102 | 62/102 | 35/101 | 17/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fixed Dose Combination (N=102) | Monotherapy Obicetrapib (N=102) | Monotherapy Ezetimibe (N=101) | Placebo (N=102)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fixed Dose Combination (N=102) | Monotherapy Obicetrapib (N=102) | Monotherapy Ezetimibe (N=101) | Placebo (N=102)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 4 (4) | 3 (3) | 3 (3)
COVID-19 (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 2 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (8) | 5 (6) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 3 (3) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (5) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 6 (6) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 4 (5) | 9 (10) | 2 (2) | 3 (3)
Fatigue (General disorders) | 4 (4) | 5 (6) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the multicenter publication or 12 months after completion of the study, whichever occurs first, Institution may publish the results of its study data. Institution and PI shall provide sponsor with an advance copy of any proposed communications at least 60 days prior and Sponsor shall have 60 days to review. Sponsor may request (a) the deletion of any Confidential Information, (b) reasonable changes, or (c) a delay for an additional period, not to exceed 90 days.

DOCUMENTS (2):
  • Study Protocol (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT06005597/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT06005597/SAP_001.pdf